CLINICAL TRIAL: NCT00938197
Title: An Open-label, Multiple-dosing, and Crossover Study to Evaluate the Pharmacokinetic Drug Interaction After Oral Concurrent Administration of Fimasartan and Amlodipine in Healthy Male Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetic Drug Interaction After Oral Concurrent Administration of Fimasartan and Amlodipine in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Choi, Director, Boryung Pharmaceutical Co., Ltd
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: A657-BR-CT-107
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Essential Hypertension
Keywords: Fimasartan; Drug interaction
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Active Comparator)
  Interventions: Drug: Fimasartan
- Part B (Active Comparator)
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Fimasartan — Fimasartan (1d~7d) Amlodipine (12d~14d) Fimasartan + Amlodipine(15d~21d)
  Arms: Part A
Drug: Amlodipine — Amlodipine (1d~10d) Amlodipine (25d~27d) Fimasartan + Amlodipine(28d~34d)
  Arms: Part B

SUMMARY:
To evaluate the pharmacokinetic drug interaction after oral concurrent administration of fimasartan and amlodipine in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* age: 20 - 40 years
* sex: male
* body weight: greater than 55 kg
* written informed consent

Exclusion Criteria:

* known allergy to Fimasartan and amlodipine
* existing cardiac or hematological diseases
* existing hepatic and renal diseases
* existing gastrointestinal diseases
* acute or chronic diseases which could affect drug absorption or metabolism
* history of any serious psychological disorder
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day 3 month ago
* participation in a clinical trial during the last 2 months prior to the start of the study

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
AUCss, Cmax,ss, Tmax,ss, CLss/F | Part A: 0, 0.5, 1, 1.5, 2, 2.5 3, 4, 6, 8, 12, 24 hours at 7 day and 21 day Part B: 0, 1, 3, 4, 5, 6, 7, 8, 9, 11, 13, 15, 24 hours at 10 day and 34 day

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Yi S, Kim TE, Yoon SH, Cho JY, Shin SG, Jang IJ, Yu KS. Pharmacokinetic interaction of fimasartan, a new angiotensin II receptor antagonist, with amlodipine in healthy volunteers. J Cardiovasc Pharmacol. 2011 Jun;57(6):682-9. doi: 10.1097/FJC.0b013e31821795d0. PMID 21394036